CLINICAL TRIAL: NCT00566501
Title: Open-Label Extension Study of 23 mg Donepezil SR in Patients With Moderate to Severe Alzheimer's Disease
Brief Title: Open-Label Extension Study of 23 mg Donepezil SR in Participants With Moderate to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2020-G000-328; 2006-004890-93 (EudraCT Number)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2021-10

CONDITIONS: Alzheimer's Disease
Keywords: Moderate-to-severe; Alzheimer's; Disease
MeSH Terms: conditions — Alzheimer Disease; Disease | interventions — Donepezil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) (Experimental): Donepezil SR 23 mg once daily orally for 12 months to participants who received donepezil 23 mg SR in the preceding double-blind study E2020-G000-326 (NCT00478205).
  Interventions: Drug: Donepezil
- Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205) (Experimental): Donepezil SR 23 mg once daily orally for 12 months to participants who received donepezil 10 mg immediate release (IR) in the preceding double-blind study E2020-G000-326 (NCT00478205).
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil SR 23 mg once daily orally.
  Other Names: Aricept

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of long-term administration of 23 milligram (mg) donepezil sustained release (SR) in participants with moderate to severe Alzheimer's disease. Participants who complete study E2020-G000-326 (NCT00478205) with no ongoing serious adverse events (SAEs) and no serious adverse drug reactions will be eligible to enter the open-label extension study.

ELIGIBILITY:
Inclusion Criteria for Participants:

1. Written informed consent from the participant (if possible) or from the participant's legal guardian or other representative at the time of the Baseline visit, prior to beginning any assessments or activities.
2. Completion of study E2020-G000-326 (NCT00478205) without ongoing SAEs or history of serious adverse drug reactions during study E2020-G000-326 (NCT00478205).
3. Participant must enroll in the present study within 3 days of completion of study E2020-G000-326 (NCT00478205).
4. Health: physically healthy and ambulatory or ambulatory-aided (that is, walker or cane); corrected vision and hearing sufficient for compliance with testing procedures.
5. Co-morbid medical conditions must be well-controlled as determined by the investigator.
6. Participants undergoing treatment with selective serotonin reuptake inhibitors (SSRIs) may be included, provided that doses are within the approved dose range as specified in the Physician's Desk Reference or local equivalent
7. Concomitant Medications: Participants undergoing treatment with the following medications may be enrolled in the study provided the following conditions are met: chronic daily benzodiazepine use if doses are stable within an approved dose range; bronchodilator medications for treatment of chronic obstructive pulmonary disease (COPD) as long as drug is administered via metered dose inhaler within approved dose range; memantine if taken at doses of 20 mg/day or less, provided that the dose is stable.
8. The participants must have a relative/caregiver who supervises the regular taking of the drug at the correct dose and is alert for possible side effects, unless the participant's legal guardian takes on this task.

Inclusion Criteria for Caregivers. Written informed consent will be obtained from the designated caregiver for participation in study assessments. The caregiver must be sufficiently familiar with the participant (as determined by the investigator) to provide accurate data. Specifically, the caregiver must have sufficient contact with the participant to provide accurate reports of the participant's functioning, must be able to observe for possible adverse events, and must be able to accompany the participant to all visits. It is preferable that the caregiver be the same as in study E2020-G000-326 (NCT00478205). If no replacement caregiver is available who meets the caregiver inclusion/exclusion criteria, the participant must be discontinued from the study.

Exclusion Criteria for Participants:

1. No caregiver available to meet the inclusion criteria for caregivers.
2. Participants with any active or clinically-significant conditions affecting absorption, distribution, or metabolism of the study medication (example, inflammatory bowel disease, gastric or duodenal ulcers, hepatic disease, or severe lactose intolerance).
3. Known plan for elective surgery during the study period that would require general anesthesia and administration of neuromuscular blocking agents, such as succinylcholine, to induce paralysis/muscle relaxation. Minor surgery, such as colonoscopy or cataract surgery, will be permitted as long as it does not require the use of these paralytic agents.
4. Participants who are unwilling or unable to fulfill the requirements of the study.
5. Use of any prohibited prior or concomitant medications.
6. Any condition that would make the participant, in the opinion of the investigator, unsuitable for the study.
7. Participant taking concomitant antidepressant medication known to have significant anticholinergic effects, such as tricyclic antidepressants prescribed at doses recommended for the treatment of major depression.
8. Participants who cannot swallow or who have difficulty swallowing whole tablets.
9. Participants taking any alternative medication such as vitamins and/or herbal products or alternative medical techniques such as acupuncture or acupressure specifically for the treatment of Alzheimer's disease.

Exclusion Criteria for Caregivers.

1. Caregivers who are unwilling or unable to give informed consent or otherwise to fulfill the requirements of the study.
2. Any condition that would make the caregiver, in the opinion of the investigator, unsuitable for the study.

Ages: 45 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2007-12-14 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Yardley, Ph.D, Study Director — Eisai Limited
Locations (1):
- Apex Research Institute, Santa Ana, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 179 centers in Asia, Europe, North America, Oceania, South Africa, and South America during 14 December 2007 to 01 April 2010. This study E2020-G000-328 (NCT00566501) was a 12-month, open-label extension of study E2020-G000-326 (NCT00478205). Participants who had received donepezil 10 milligram (mg) immediate release (IR) or donepezil 23 mg sustained release (SR) during Study E2020-G000-326 (NCT00478205) were eligible for enrollment into this study.
Pre-assignment Details: A total of 1084 participants completed the study E2020-G000-326 (NCT00478205), of which 915 participants were enrolled and signed informed consent form and out of them, 902 participants received treatment in this study E2020-G000-328 (NCT00566501).
Groups:
- Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205): Donepezil SR 23 mg once daily orally for 12 months to participants who received donepezil 10 mg IR in the preceding double-blind study E2020-G000-326 (NCT00478205).
Period: Overall Study
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Started | 570 | 332
Completed | 423 | 210
Not Completed | 147 | 122
Not completed — Adverse Event | 68 | 59
Not completed — Medication Non-compliance | 5 | 0
Not completed — Protocol Violation | 2 | 2
Not completed — Request of Investigator or Sponsor | 6 | 7
Not completed — Withdrawal by Subject | 33 | 30
Not completed — Lack of Efficacy | 8 | 3
Not completed — Other | 25 | 21

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least one dose of the study medication during the open-label treatment period and had at least one post-baseline safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205) | Total
Number analyzed (Participants) | 570 | 332 | 902
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (8.67) | 74.5 (8.44) | 74.3 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 373 | 202 | 575
  Male | 197 | 130 | 327
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 16 | 7 | 23
  White | 429 | 245 | 674
  Hispanic | 42 | 18 | 60
  Asian/Pacific | 80 | 60 | 140
  Other | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product, whether or not considered related to the investigational product, a change in treatment, or discontinuation of study drug, recurrence of an intermittent medical condition not present pretreatment, an abnormal laboratory test result was considered an AE if the identified laboratory abnormality led to any type of intervention, withdrawal of study drug, or withholding of study drug, whether prescribed in the protocol or not. All AEs in Study 328 (NCT00566501) excluding treatment-emergent signs or symptoms continuing from Study 326 (NCT00478205) were reported.
Time Frame: From the enrollment of the study up to 30 days after last dose of the study drug (up to 2 years 3 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 570 | 332
Participants | 416 | 259

2. Secondary Outcome: Percentage of Participants With at Least 1 Treatment-Emergent Abnormal Laboratory Values (TEAVs): Hematology
Description: A TEAV for a laboratory parameter was defined as a value that was clinically significantly outside (above or below) the normal range post-dose, but within the normal range prior to drug administration, or a value that represented a clinically significant exacerbation of an abnormality present prior to drug administration. Abnormal values for hematology parameters were: White Blood cells count: less than or equal to [<=] 2,800/per millimeter (mm) or greater than or equal to [>=] 16,000/mm; Neutrophils: <=15 percent (%); Hemoglobin: Male (<=11.5 gram per deciliter [g/dL]), Female (<=9.5 g/dL); Hematocrit: Male (<=37%), Female (<=32%); Eosinophils: >=10%; Platelet Count: <=75,000/mm or >=700,000/mm. Percentage of participants with at least 1 abnormal TEAV for hematology was reported.
Time Frame: From the first dose of study drug up to 2 years 3 months
Population: The safety population included all participants who received at least one dose of the study medication during the open-label treatment period and had at least one post-baseline safety assessment. Here 'N' (overall number analyzed) are the participants who were evaluable for the outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 546 | 311
percentage of participants | 9.5 | 10.9

3. Secondary Outcome: Percentage of Participants With at Least 1 TEAVs for Selected Parameters: Clinical Chemistry
Description: A TEAV for a laboratory parameter was defined as a value that was clinically significantly outside (above or below) the normal range postdose, but within the normal range prior to drug administration,or a value that represented a clinically significant exacerbation of an abnormality present prior to drug administration.Abnormal values for clinical chemistry parameters were:Sodium:Less than(<)130 milliequivalents per litre (mEq/L) or greater than(>)150 mEq/L;Potassium:<3 mEq/L or >5.5 mEq/L; Calcium: <8.4 milligram per deciliter (mg/dL) or >1.5 mg/dL;Albumin: 50% lower limit of normal (LLN); Alkaline Phosphatase:>=3*upper limit of normal (ULN);Aspartate aminotransferase (AST):>=3*ULN;Alanine aminotransferase(ALT):>=3*ULN;Total Bilirubin:>=2.0 mg/dL;Chloride:<90 mEq/L or >115 mEq/L;Creatinine:>=2.0 mg/dL;Creatine phosphokinase:>=3*ULN;Blood Urea Nitrogen (BUN):>=30 mg/dL. Percentage of participants with at least 1 abnormal TEAV (selected parameters) for clinical chemistry was reported.
Time Frame: From the first dose of study drug up to 2 years 3 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 553 | 312
percentage of participants | 14.3 | 13.1

4. Secondary Outcome: Change From Baseline in Severe Impairment Battery (SIB) Total Score
Description: The SIB evaluated the severity of cognitive dysfunction in participants with more advanced dementia. Test questions measured attention, language, orientation, memory, praxis, visuospatial ability, construction, social skills, orienting head to name. Non-verbal responses were allowed, thus decreasing the need for language output. Forty questions were included with a total possible score range of 0-100. Lower scores indicated greater cognitive impairment.
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: The Intent-to-treat (ITT) population included all safety participants who have at least one post-baseline efficacy measurement. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure and 'n' (number analyzed) included all participants who were evaluable at specified timepoints for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 546 | 311
score on a scale
  At Baseline | 78.4 (19.05) | 77.2 (19.49)
  Change at Month 3: number analyzed (Participants) | 546 | 309
  Change at Month 3 | -1.7 (7.11) | -0.9 (6.55)
  Change at Month 6: number analyzed (Participants) | 492 | 270
  Change at Month 6 | -4.0 (9.52) | -2.8 (8.68)
  Change at Month 9: number analyzed (Participants) | 462 | 239
  Change at Month 9 | -5.5 (11.19) | -5.2 (9.71)
  Change at Month 12: number analyzed (Participants) | 423 | 207
  Change at Month 12 | -7.5 (12.99) | -6.7 (10.75)

5. Secondary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Total Score
Description: MMSE is a 30-point scale that measured orientation to time and place, registration, immediate and delayed recall, attention, language, and drawing. Scores ranged from 0 (most impaired) to 30 (no impairment). Lower score indicated more impairment.
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: The ITT population included all safety participants who have at least one post-baseline efficacy measurement. Here 'N' (overall number of participants analyzed) included all participants who were evaluable for this outcome measure and 'n' (number analyzed) included all participants who were evaluable at specified timepoints for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 549 | 314
score on a scale
  Baseline | 14.1 (5.81) | 13.8 (6.02)
  Change at Month 3: number analyzed (Participants) | 547 | 314
  Change at Month 3 | -0.6 (2.27) | -0.5 (2.20)
  Change at Month 6: number analyzed (Participants) | 493 | 270
  Change at Month 6 | -1.3 (2.70) | -1.2 (2.53)
  Change at Month 9: number analyzed (Participants) | 468 | 240
  Change at Month 9 | -1.7 (2.95) | -1.7 (2.77)
  Change at Month 12: number analyzed (Participants) | 428 | 208
  Change at Month 12 | -2.3 (3.08) | -2.1 (3.04)

6. Secondary Outcome: Change From Baseline in Modified Alzheimer's Disease Cooperative Study Activities of Daily Living Severe Scale (ADCS-ADL) Total Score
Description: ADCS-ADL is a comprehensive battery of ADL questions used to measure a participant's functional capabilities. The modified ADCS-ADL-severe scale is a 19-item scale that has been validated for the assessment of participants with moderate to severe dementia. It measured the most appropriate basic and instrumental abilities (such as walking, grooming, bathing, and eating) in this participant population. Response to each item was obtained by interview with the caregiver. Ratings reflected caregiver observations about the participant's actual functioning and provided an assessment of change in the functional state of the participant over time. The total score ranged from 0 to 54. Lower scores indicated greater functional impairment.
Time Frame: At Baseline, Month 3, Month 6, Month 9 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 556 | 315
score on a scale
  Baseline | 34.3 (11.26) | 34.3 (11.26)
  Change at Month 3: number analyzed (Participants) | 555 | 315
  Change at Month 3 | -1.6 (5.30) | -1.8 (5.27)
  Change at Month 6: number analyzed (Participants) | 500 | 273
  Change at Month 6 | -3.2 (6.13) | -3.7 (6.53)
  Change at Month 9: number analyzed (Participants) | 471 | 245
  Change at Month 9 | -4.6 (6.91) | -4.8 (7.46)
  Change at Month 12: number analyzed (Participants) | 433 | 213
  Change at Month 12 | -5.6 (7.62) | -6.8 (8.96)

7. Secondary Outcome: Change From Baseline in Quality of Life-Alzheimer's Disease (Qol-AD) Total Score
Description: QoL-AD is a 13-item quality of life instrument developed to specifically assess QoL in participants who have dementia. Each item was scored on a 4-point scale (poor, fair, good, excellent) and a single score was calculated, ranging from 13 (low functioning) to 52 (normal function). Higher score indicated better QoL. The QoL-AD total scores for the participants and caregiver were the sum of the 13 items on each test.
Time Frame: At Baseline, Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 527 | 301
score on a scale
  Caregiver; Baseline | 31.6 (6.37) | 30.8 (6.62)
  Caregiver; Change at Month 6: number analyzed (Participants) | 525 | 299
  Caregiver; Change at Month 6 | -1.4 (5.17) | -1.4 (5.08)
  Caregiver; Change at Month 12: number analyzed (Participants) | 437 | 219
  Caregiver; Change at Month 12 | -1.8 (5.60) | -1.8 (5.28)
  Participant; Baseline: number analyzed (Participants) | 465 | 271
  Participant; Baseline | 35.2 (6.65) | 34.5 (6.90)
  Participant; Change at Month 6: number analyzed (Participants) | 453 | 266
  Participant; Change at Month 6 | -0.2 (5.10) | -0.1 (4.95)
  Participant; Change at Month 12: number analyzed (Participants) | 376 | 187
  Participant; Change at Month 12 | -0.2 (5.02) | -0.2 (4.76)

8. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimension (EQ-5D) Total Score
Description: EQ-5D is a health profile questionnaire assessing quality of life along 5 domains. Caregivers rated 5 domains of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) by choosing from 3 answering options (1=no problems; 2=some problems; 3=extreme problems). The EQ-5D Health Utilities Index (HUI) is derived from the five dimensions of the EQ-5D, using country-specific preference weights (tariffs) to summarize how good or bad each health state is on a scale from 1 to 0. HSI total score ranged from 1 (full health) and 0 (worst health/death).
Time Frame: At Baseline, Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 531 | 303
score on a scale
  Baseline | 0.76 (0.17) | 0.77 (0.19)
  Change at Month 6: number analyzed (Participants) | 530 | 303
  Change at Month 6 | -0.04 (0.15) | -0.04 (0.18)
  Change at Month 12: number analyzed (Participants) | 437 | 217
  Change at Month 12 | -0.06 (0.18) | -0.06 (0.19)

9. Secondary Outcome: Change From Baseline in Screen for Caregiver Objective Burden (SCB) Total Score
Description: The SCB is a 25-item instrument that questions caregivers about the occurrence and degree of distress as aspects of the burden of care during the preceding two weeks. It was designed specifically for use with caregivers of Alzheimer's disease participants. Each item was assessed on a 5-point scale ranging from "0" (no occurrence) to "4" (occurrence with severe distress). The objective burden was the sum of the total numbers of (1 2 3 4) in all items. Total score ranged from 0 (low distress) to 100 (high distress).
Time Frame: At Baseline, Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 520 | 296
score on a scale
  Baseline | 9.8 (4.36) | 9.8 (4.74)
  Change at Month 6: number analyzed (Participants) | 516 | 295
  Change at Month 6 | 0.5 (3.76) | 1.0 (3.64)
  Change at Month 12: number analyzed (Participants) | 430 | 216
  Change at Month 12 | 1.2 (3.94) | 1.5 (3.98)

10. Secondary Outcome: Change From Baseline in Screen for Caregiver Subjective Burden (SCB) Total Score
Description: The SCB is a 25-item instrument that questioned caregivers about the occurrence and degree of distress as aspects of the burden of care during the preceding two weeks. It was designed specifically for use with caregivers of Alzheimer's disease participants. Each item was assessed on a 5-point scale ranging from "0" (no occurrence) to "4" (occurrence with severe distress). The subjective burden was the sum of the (total number with score*score). Total score ranged from 0 (no occurrence) to 100 (occurrence with severe distress).
Time Frame: At Baseline, Month 6 and Month 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 520 | 296
score on a scale
  Baseline | 18.4 (10.98) | 18.5 (12.14)
  Change at Month 6: number analyzed (Participants) | 516 | 295
  Change at Month 6 | 1.7 (10.03) | 3.0 (9.63)
  Change at Month 12: number analyzed (Participants) | 430 | 216
  Change at Month 12 | 3.2 (10.30) | 4.3 (10.64)

11. Secondary Outcome: Number of Participants With Treatment Outcome Scale (TOS) Score
Description: TOS is a pilot instrument designed to evaluate the caregiver's assessment of the participant's status. The caregiver was asked how much he/she thinks the participant has been helped by participating in the study. This instrument comprised a 7-point Likert scale in which a rating of 1=Very much improved; 2=Moderately improved; 3=Minimally improved; 4=About the same; 5=Minimally worse; 6=Moderately worse; 7=Very much worse. The total scale ranged from 1 (marked improvement) to 7 (marked worsening).
Time Frame: At Months 6 and 12
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 530 | 302
Participants
  At Month 6: 1=Very much improved | 10 | 7
  At Month 6: 2=Moderately improved | 56 | 29
  At Month 6: 3=Minimally improved | 66 | 40
  At Month 6: 4=About the same | 149 | 79
  At Month 6: 5=Minimally worse | 130 | 73
  At Month 6: 6=Moderately worse | 96 | 57
  At Month 6: 7=Very much worse | 23 | 17
  At Month 12: number analyzed (Participants) | 440 | 222
  At Month 12: 1=Very much improved | 12 | 5
  At Month 12: 2=Moderately improved | 37 | 20
  At Month 12: 3=Minimally improved | 67 | 23
  At Month 12: 4=About the same | 91 | 52
  At Month 12: 5=Minimally worse | 103 | 42
  At Month 12: 6=Moderately worse | 89 | 54
  At Month 12: 7=Very much worse | 41 | 26

12. Secondary Outcome: Goal Attainment Scaling (GAtS) Score Total Score
Description: GAtS is a technique that is standardized with respect to the general approach, but individualized with respect to the outcome goals of each participant. GAtS was designed to provide insight into the changes that are considered as important by the caregiver and (if feasible) by the participants. At study initiation, the participants (if capable) and, separately, the caregiver were asked to specify up to 4 goals for the participants during study participation. For each goal, a description of the current state (or one supplied with the help of the clinician if necessary) was provided to anchor the baseline assessment at 0, and other possible outcomes were described. The outcome for each goal was quantified by a 4-point scale that provided for improvement (+1, +2), no change (0) or worsening (-1, -2). Total score ranged from -30 (worsened) to 130 (most improved). Baseline score was set to be 50 (when scores of all goals are '0' [no change]).
Time Frame: At Months 6 and 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
Number analyzed (Participants) | 510 | 295
score on a scale
  Caregivers; At Month 6: number analyzed (Participants) | 505 | 291
  Caregivers; At Month 6 | -2.6 (9.63) | -3.2 (9.97)
  Caregivers At Month 12: number analyzed (Participants) | 423 | 213
  Caregivers At Month 12 | -5.1 (11.10) | -5.9 (10.61)
  Participants; At Month 6: number analyzed (Participants) | 107 | 67
  Participants; At Month 6 | 2.2 (7.34) | -0.8 (8.26)
  Participants; At Month 12: number analyzed (Participants) | 95 | 49
  Participants; At Month 12 | 2.4 (7.89) | -0.6 (9.57)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 2 years 3 months
Arm/Group | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205)
All-Cause Mortality (participants affected / at risk) | 14/570 | 5/332
Serious Adverse Events (participants affected / at risk) | 80/570 | 56/332
Other Adverse Events (participants affected / at risk) | 415/570 | 259/332
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) (N=570) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205) (N=332)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Encephalocele (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Meningocele (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 2 | 0
Gait disturbance (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Orchitis (Infections and infestations) | 1 | 0
Peritonillar abscess (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 6 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 8 | 3
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Device lead damage (Injury, poisoning and procedural complications) | 1 | 0
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 7 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Lipase increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradykinesia (Nervous system disorders) | 0 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrospinal fistula (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 5 | 2
Convulsion (Nervous system disorders) | 1 | 0
Dementia Alzheimers type (Nervous system disorders) | 2 (570) | 0
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Ischemic cerebral infarction (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 6 | 6
Transient ischemic attack (Nervous system disorders) | 1 | 3
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 3
Agitation (Psychiatric disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 3
Mental status change (Psychiatric disorders) | 0 | 4
Poriomania (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Cardio-rspiratory arrest (Cardiac disorders) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil SR 23 mg (Donepezil SR 23 mg in Study NCT00478205) (N=570) | Donepezil SR 23 mg (Donepezil IR 10 mg in Study NCT00478205) (N=332)
Weight decreased (Investigations) | 58 | 43
Fall (Injury, poisoning and procedural complications) | 54 | 25
Agitation (Psychiatric disorders) | 33 | 28
Urinary tract infection (Renal and urinary disorders) | 33 | 20
Diarrhoea (Gastrointestinal disorders) | 20 | 19
Aggression (Psychiatric disorders) | 29 | 23
Nausea (General disorders) | 12 | 20
Insomnia (Gastrointestinal disorders) | 18 | 15
Hypertension (Vascular disorders) | 18 | 10
Syncope (Nervous system disorders) | 19 | 9
Depression (Psychiatric disorders) | 15 | 12
Weight increased (Investigations) | 15 | 12
Nasopharyngitis (Infections and infestations) | 14 | 11
Vomiting (Gastrointestinal disorders) | 9 | 15
Urinary incontinence (Renal and urinary disorders) | 12 | 11
Anorexia (Metabolism and nutrition disorders) | 11 | 11
Irritability (General disorders) | 13 | 7
Oedema peripheral (General disorders) | 15 | 5
Asthenia (General disorders) | 6 | 12
Dizziness (Nervous system disorders) | 6 | 12
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 7
Contusion (Injury, poisoning and procedural complications) | 9 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8
Anxiety (Psychiatric disorders) | 12 | 2
Constipation (Gastrointestinal disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Anaemia (Blood and lymphatic system disorders) | 3 | 9
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Haematuria (Renal and urinary disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No